CLINICAL TRIAL: NCT05549557
Title: An Open-label, Multi-center Phase I Clinical Study of IMM40H in Patients With Advanced Solid Tumor and Hematological Malignancies
Brief Title: IMM40H Phase I Dose Escalation and Expansion
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ImmuneOnco Biopharmaceuticals (Shanghai) Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMM40H-01
Record Dates: First submitted 2022-09-15; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IMM40H (Experimental): IMM40H is a monoclonal antibody with target CD70.
  Interventions: Drug: IMM40H

INTERVENTIONS:
Drug: IMM40H — IMM40H is a monoclonal antibody with a molecular generated from ImmuneOnco's antibody platform. IMM40H targets CD70 (a tumor cell marker).
  Other Names: study drug: IMM40H

SUMMARY:
This is first-in-human, open-label, multi-center, dose-escalation (phase Ia) and cohort expansion (phase Ib) phase I study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamic, immunogenicity, and antitumor activities of IMM40H in patients with advanced malignancies including solid tumor and hematological malignancies.

DETAILED DESCRIPTION:
This study will include 16~27 patients with advanced malignancies that have progressed after or have no response to previous standard treatments or for whom no standard treatments are available (including but not limited to melanoma, nasopharyngeal cancer, thymoma, RCC, colorectal cancer, non-small cell lung cancer (NSCLC), glioblastoma, astrocytoma, ovarian cancer, AML, and lymphoma). The primary objective is to determine the maximum tolerated dosage (MTD) or recommended dose for expansion (RDE) by observing the safety and tolerability of IMM40H monotherapy.

The adjusted "3 + 3" design will be adopted in this trial for dose escalation, with the starting dose of IMM40H at 0.3 mg/kg and the temporary maximum dose at 20 mg/kg. In the dose-escalation stage, a total of 5 dose levels will be designed:0.3, 1, 3, 10, 20 mg/kg, to determine MTD . For each subject in each dose group, the dose will be gradually increased according to the dose-escalation rules, and the observation period for dose-limiting toxicity (DLT) will be set to be 28 days after the first dose.

Patients with CD70-positive malignancies to further evaluate the safety, PK characteristics, immunogenicity, and anti-tumor activity or preliminary efficacy of IMM40H dosing at MTD.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old; no gender limitation;
2. Expected survival time ≥12 weeks;
3. ECOG score is 0 - 1 points;
4. The interval between the first dose of previous anti-tumor therapy and the first dose must meet the following conditions:

1)Subjects who have received chemical drugs, small molecule targeted therapy drugs, immunomodulators or Chinese patent medicines with clear anti-tumor indications in the past should discontinue the drug for at least 2 weeks or 5 half-lives, whichever is shorter; 2)Subjects who have received macromolecular targeted drugs and protein preparations in the past should discontinue the drug for 5 half-lives or 4 weeks, whichever is shorter; 3)Subjects who have previously received radiotherapy, cell transplantation, CAR-T or immune checkpoint inhibitors such as PD-1/PD-L1 therapy should discontinue the drug for at least 4 weeks; 5. Subjects who have suitable organ function and hematopoietic function:

1. Neutrophil count ≥1.0 × 109/L; (no short-acting drugs for leucopenia within 1 week; no long-acting drugs for leucopenia within 3 weeks, such as granulocyte colony-stimulating factor);
2. Platelet count ≥75 × 109/L (without bone marrow infiltration) / ≥50 × 109/L (with bone marrow infiltration); (have not received platelet transfusion therapy within 1 week);
3. Hemoglobin ≥80 g/L (without bone marrow infiltration) / ≥70 g/L (with bone marrow infiltration); (have not received red blood cell transfusion therapy or biological response modifiers such as erythropoietin within 2 weeks);
4. Total bilirubin (TBIL) ≤ 1.5 × ULN; TBIL ≤ 3 × ULN if there is liver metastasis;
5. Both aspartate aminotransferase (AST) and alanine aminotransferase (ALT) should be ≤2.5×ULN; if there is liver metastasis, both AST and ALT should be ≤5.0×ULN;
6. International normalized ratio (INR) ≤ 2 × ULN, or activated partial thromboplastin time (APTT) ≤ 2.0 × ULN;
7. Heart: left ventricular ejection fraction (LVEF) ≥ 50%;
8. Creatinine clearance (CrCl) ≥30 mL/min/1.73m2 or serum creatinine (Cr) ≤1.5 × ULN; 6. Subjects who have AEs related to previous systemic chemotherapy, radical/extensive radiotherapy or other anti-tumor drug treatment recovered to (NCI CTCAE v5.0) ≤ grade 1 (except for alopecia, skin hyperpigmentation, skin induration, skin atrophy, which are not clinically significant or those with no clinical significance in the opinion of the investigator); 7. Men and women of childbearing age should agree to take effective contraceptive measures such as barrier contraception, hormonal contraception or long-term use of contraceptives from the time of signing the informed consent to 3 months after the last dose.

8. Subjects should voluntarily sign the informed consent form, understand the study and be willing to follow the protocol requirements and have the ability to complete all experimental procedures.

9. Subjects' diseases can be assessed.

Exclusion Criteria:

1. Subjects have received CD70-targeted therapy in the past; 2. Subjects who have received allogeneic transplantation in the past and require continuous use of immunosuppressive agents; 3. Patients who have primary central nervous system (CNS) malignant tumor or patients with active CNS metastases who have failed local treatment (radiotherapy or surgery), but the following patients are allowed to be enrolled: a. asymptomatic brain metastases; b. clinically stable (i.e. no imaging progression was seen 4 weeks before the first dose, and any neurological symptoms had returned to baseline levels) and no treatment for brain metastases was required; 4. Subjects who have serious organic disease, or the investigator judges that it is not suitable to participate in the study due to the combination of other serious diseases:

1. Have hypertension, pulmonary hypertension, or unstable angina that is difficult to control with medication;
2. Have myocardial infarction or bypass or stent surgery within 6 months before administration;
3. History of chronic heart failure with New York Heart Association (NYHA) criteria 3-4 within 6 months prior to administration;
4. Have serious arrhythmias requiring treatment (excluding atrial fibrillation, polymorphic ventricular tachycardia), including QTc ≥450ms for men and ≥470ms for women (calculated by Fridericia formula);
5. Have cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 12 months before enrollment;
6. History of arterial thrombosis, deep vein thrombosis and pulmonary embolism within 3 months before administration;
7. History of moderate or severe dyspnea at rest, or current need for continuous oxygen therapy, or current interstitial lung disease (ILD) or pneumonia, severe chronic obstructive pulmonary disease, severe pulmonary insufficiency, symptomatic bronchospasm;
8. Presence of a disorder that may cause gastrointestinal bleeding or perforation (e.g. symptomatic duodenal ulcer requiring treatment, intestinal obstruction, acute or chronic Crohn's disease, ulcerative colitis, or those with a history of intestinal perforation and intestinal fistula who have not been cured);
9. The puncture and drainage treatment cannot control the disease and repeated drainage is required or there is pleural, abdominal or pericardial effusion with obvious symptoms; 5. Subjects who have active viral hepatitis B (HBsAg positive and/or HBcAb positive, and HBV DNA ≥1000 IU/mL), or active viral hepatitis C (anti-HCV antibody positive, and HCV RNA higher than the lower limit), or who are HIV-infected.

6. Subjects who have active autoimmune disorders and need to rely on immunosuppressive therapy or receive systemic hormone therapy with a dose of ≥10 mg/day of prednisone or other equivalent hormones within 2 weeks before enrollment; 7. Subjects who have uncontrollable serious active infection (such as sepsis, bacteremia, viremia, etc.); 8. Subjects who have received live attenuated vaccine within 4 weeks before the first administration; 9. Subjects who have major surgery within 4 weeks before the first administration or plan to take major surgery within 3 months after the first administration of the study drug, excluding intubation, peripheral venipuncture, central venous catheterization, etc.; 10. Subjects who have a history of neurological or mental disorders and have been hospitalized within the past six months, and have a history of alcohol and drug abuse within the past year; 11. Women with positive serum pregnancy test or during the lactation period; 12. Men and women of childbearing age are unwilling to take adequate contraceptive measures during the study period and within 3 months after the last dose; 13. Other circumstances that the investigator considers inappropriate to participate in this study.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of IMM40H in patients with advanced malignancies. | 28 days
  DLT

SECONDARY OUTCOMES:
To evaluate the maximum observed plasma concentration (Cmax) of IMM40H in patients with advanced malignancies; | 6 months
  maximum observed plasma concentration (Cmax) characteristics
To evaluate the time at which Cmax occurred (Tmax) of IMM40H in patients with advanced malignancies; | 6 months
  the time at which Cmax occurred (Tmax) characteristics
To evaluate the area under the plasma drug concentration-time curve from time 0 to the last quantifiable time point (AUC0-t) of IMM40H in patients with advanced malignancies; | 6 months
  the area under the plasma drug concentration-time curve from time 0 to the last quantifiable time point (AUC0-t) characteristics
To evaluate the area under the plasma drug concentration-time curve from time 0 extrapolated to infinity (AUC0-∞) of IMM40H in patients with advanced malignancies; | 6 months
  the area under the plasma drug concentration-time curve from time 0 extrapolated to infinity (AUC0-∞) characteristics
To evaluate the terminal half-life (t1/2) of IMM40H in patients with advanced malignancies; | 6 months
  the terminal half-life (t1/2) characteristics

OTHER OUTCOMES:
To explore the potential biomarker for IMM40H therapy; | 6 months
  CD70 and sCD27 express

IPD SHARING:
Plan to Share IPD: No